CLINICAL TRIAL: NCT05237531
Title: Preop Education and Opioid Use After Hand and Wrist Fracture ORIF: A Randomized Controlled Trial at a County Hospital
Brief Title: Preoperative Education in Hand and Wrist Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty enrolling participants.
Sponsor: Emory University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Principal Investigator, Paul A Ghareeb, MD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003074
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Distal Radius Fracture
Keywords: ORIF
MeSH Terms: conditions — Wrist Fractures | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Patients in the experimental arm will receive standardized preoperative education in the form of a brief video, interactive quiz, and written handout.
  All patients will receive standardized multimodal pain management consisting of a long-acting peripheral nerve block, scheduled non-opioid pain medications, an opioid prescription to be taken only as needed, and adjunctive medicines to be taken as needed for any side effects.
  Interventions: Behavioral: Standardized Preoperative Education; Behavioral: Preoperative and postoperative questionnaires
- Control Arm (Active Comparator): Patients in the control arm will receive education per the provider's preference (current standard of care).
  All patients will receive standardized multimodal pain management consisting of a long-acting peripheral nerve block, scheduled non-opioid pain medications, an opioid prescription to be taken only as needed, and adjunctive medicines to be taken as needed for any side effects.
  Interventions: Behavioral: Standard of care; Behavioral: Preoperative and postoperative questionnaires

INTERVENTIONS:
Behavioral: Standardized Preoperative Education — The standardized preoperative education includes a brief video, an interactive quiz, and a written handout.
  The video will provide information on the proper use and common side effects of opioid pain medications, the expected effects of a peripheral nerve block, and the concept of multimodal postoperative pain management with non-opioid medications and non-pharmaceutical pain management strategies. The interactive quiz will reinforce the critical components of the video in a question-and-answer format which requires active participation. The written handout will summarize the educational content in a form which can be easily referenced by patients at home.
  Arms: Experimental Arm
Behavioral: Standard of care — Education per provider preference (no standardization, current standard of care)
  Arms: Control Arm
Behavioral: Preoperative and postoperative questionnaires — Preoperative questionnaire: Demographic questions plus specific questions about chronic pain, prior opioid use, and mental health diagnoses Postoperative questionnaire: Questions about pain control after surgery, satisfaction with pain control, healthcare contact since surgery, opioid consumption since surgery, and satisfaction with education

SUMMARY:
This study will compare opioid consumption in patients undergoing outpatient surgical fixation of distal radius fractures with and without standardized preoperative education at Grady Memorial Hospital.

DETAILED DESCRIPTION:
The proposed research aims to study the impact of preoperative education on postoperative pain control after outpatient surgery for traumatic wrist fractures. The impact of preoperative education will be studied through patient questionnaires and by tracking postoperative opioid consumption as well as instances of unscheduled healthcare contact after surgery. The study will be a randomized controlled trial. This study imposes no more than minimal risk to study participants. Loss of privacy and breach of confidentiality are risks of this study. All data will be stored securely on Microsoft One Drive, a password-protected, encrypted database which requires two-factor authorization. The study population will be patients aged 18-99 years who are undergoing outpatient surgical management of distal radius fractures at Grady Memorial Hospital. No vulnerable populations will be included. Contact will be made with potential study participants at their preoperative clinic visit. Written informed consent will be obtained. Data will not be publicly available. Data will be deidentified, and no members of the team will have access to the code that identifies patients. Data will be collected in the plastic surgery clinic, orthopedic surgery clinic, and preoperative area at Grady Memorial Hospital. The total respondent burden will be 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 years with a closed carpal, metacarpal, or distal radius fracture undergoing outpatient surgical management at Grady Memorial Hospital, who is willing to participate and mentally capable to consent.

Exclusion Criteria:

* Patients who are inpatients at the time of surgery. Patients who have concomitant injuries on the same extremity as the carpal, metacarpal, or distal radius fracture. Patients with open fractures. Patients unable to tolerate non-steroidal anti-inflammatory drugs (NSAIDs). Non-English speaking patients will be excluded.
* Adults who are unable to consent will not be included.
* Individuals who are not yet adults will not be included.
* Pregnant women will not be included.
* Prisoners will not be included.
* Cognitively impaired individuals or individuals with impaired decision-making capacity will not be included.
* Individuals who speak English will be included. Individuals who have limited English proficiency but speak Spanish as a primary language will not be eligible for inclusion. Spanish-speaking patients will be excluded because the components of the educational protocol (video, questionnaires, surveys) are not available in Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Change in total oral morphine equivalents consumed from day of surgery to postoperative day 10 | Day of surgery, postoperative day 10
  Change in oral morphine equivalents consumed from day of surgery to postoperative day 10 (POD 10). The total amount of morphine equivalents consumed between the 2 study arms will be compared.

SECONDARY OUTCOMES:
Total opioid consumption during the postoperative course | Up to postoperative day 10
  Total opioid consumption in mg during the postoperative course taken from the pain diary and postoperative questionnaire.
Total number of opioid refills in the postoperative period | Up to postoperative day 10
  Number of opioid refills in the postoperative period based on postoperative questionnaire and prescription drug monitoring program (PDMP) database.
Change in average daily VAS pain scores for early (postoperative day 0-3), middle (postoperative day 4-7), and late (postoperative day 8-10) postoperative period between the two study arms | Baseline, postoperative day 0-3, postoperative day 4-7, postoperative day 8-10
  Average visual analog scale (VAS) pain score will be collected for early (postoperative day 0-3), middle (postoperative day 4-7), and late (postoperative day 8-10) postoperative period from the pain diary, and results will be compared between both study arms. Total score ranges between 1-10 and 10 correlates with worse pain.
Total number of unscheduled healthcare contact (UHC) up to 30 days after surgery | Up to 30 days after surgery
  UHC includes telephone calls to clinical staff (documented in electronic medical record), early clinic visits, emergency room visits, and readmissions to the hospital
Type of reason of unscheduled healthcare contact (UHC) up to 30 days after surgery | Up to 30 days after surgery
  UHC includes telephone calls to clinical staff (documented in electronic medical record), early clinic visits, emergency room visits, and readmissions to the hospital. The reason will be collected from the day of surgery until 30 days after surgery.
Change in results of Pain Management quiz after education | Preoperative, day of surgery
  Change in results of Pain Management Quiz before and after education. Answers to the questions on the quiz are either correct or incorrect. Total number questions are 11. It will be measured as total number of correct answers/total number of questions (number of correct/11). This will be converted to a percentage correct. Range of score will be 0% - 100% correct. Higher change in percentage correct is a better outcome. Change in percentage correct from preoperative appointment to day of surgery will help determine the effectiveness of the educational protocol.
Postoperative Satisfaction score with education | Postoperative (up to 2 weeks after surgery)
  Based on the postoperative questionnaire, participants will answer a question about satisfaction with 5 possible answers: Very satisfied, Somewhat satisfied, Neutral, Somewhat dissatisfied and Very dissatisfied.
  Results will be in percentage, based on number of participants in each category. "Very satisfied" correlates with better outcome with lower level of satisfaction until "very dissatisfied" that correlates with worse outcome.
Percentage of participants with adequate postoperative pain control | Postoperative (Up to 2 weeks after surgery)
  Based on the postoperative questionnaire, participants will answer a question about pain control:
  "Do you feel like your pain was adequately controlled after surgery?" Possible answers include:Yes, No and Somewhat.
  Number of participants who answer "Yes" will be counted per randomization group. A higher result correlates with better outcome (better pain control).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ghareeb, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: * Anyone who wishes to access the data
  * Any purpose
  * Data will be available indefinitely